CLINICAL TRIAL: NCT07369349
Title: Artificial Intelligence Application of Neurogenic Bowel Training in Patients With Spinal Cord Injury
Brief Title: Artificial Int: Neurogenic Bowel Education in Spinal Cord Injury Patients
Acronym: ArtInt
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Senem Duman (Other)
Responsible Party: Sponsor-Investigator, Senem Duman, Lecturer, Saglik Bilimleri Universitesi
Organization: Saglik Bilimleri Universitesi (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SaglikBilimleriU-1; Ethics Committee (Other: Ankara City Hospital Ethics Committee)
Record Dates: First submitted 2025-08-27; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injury; Neurogenic Bowel Dysfunction
Keywords: spinal cord injury; neurogenic bowel dysfunction; Artificial Intelligence
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group consisted of participants who only received the hospital's routine NBD education. No additional intervention was provided. The NBD education was delivered by clinical nurses. At the end of the 4th and 12th weeks, the links for the post-tests were sent to the participants in the control group via WhatsApp messages to their phones. After the completion of the study, a link to the mobile application was also provided to the control group via WhatsApp along with an explanatory note.
- intervention group (Experimental): İndividuals in the intervention group will receive the same routine education as the control group. In addition to the routine education, on the day of discharge, a link will be sent to their phones through which the mobile application will be downloaded. Participants will create an account in the mobile application by entering their name, surname, and password. The purpose of installing the mobile application on the day of discharge is to prevent individuals in the control group from becoming aware of the mobile application. After discharge, participants will be followed up during the 4th and 12th weeks.
  Interventions: Other: Mobil Application

INTERVENTIONS:
Other: Mobil Application — After discharge, the documents to be completed will be delivered to the intervention group participants via the mobile application and to the control group participants via WhatsApp. At the end of the study, after the final assessment is completed, participants will be informed of their group allocation, and those in the control group will be provided with access to the mobile application via a WhatsApp link.
  Arms: intervention group

SUMMARY:
The aim of this study is to evaluate the effectiveness of patient education delivered through an artificial intelligence (AI)-based mobile application in the management of neurogenic bowel dysfunction in individuals with spinal cord injury. Within the scope of the study, it will be examined whether the mobile application reduces neurogenic bowel scores, contributes to maintaining stool scores within the normal range, and improves the quality of life of individuals. Accordingly, the AI-based education model to be developed is expected to facilitate the integration of bowel management practices into daily life, prevent complications, and enhance social participation.

-

ELIGIBILITY:
Inclusion Criteria:

* Volunteers who consent to participate.
* Age over 18 years.
* Diagnosed with spinal cord injury (SCI).
* Diagnosed with neurogenic bowel dysfunction (NBD).
* Not in spinal shock (return of the bulbocavernosus reflex).
* Having received routine NBD education at the study center within the last month.

Exclusion Criteria:

* Individuals with mental retardation.
* Individuals with visual and/or hearing impairments.
* Individuals with communication problems.
* Individuals with a history of additional injuries other than SCI (e.g., head trauma, pelvic injury, pelvic surgery).
* Individuals diagnosed with neurological disorders such as stroke, Parkinson's disease, polyneuropathy, or multiple sclerosis.
* Individuals with irritable bowel syndrome (IBS) or inflammatory bowel disease (IBD).
* Individuals diagnosed with gastrointestinal malignancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Neurogenic Bowel Dysfunction (NBD) Score Assessed by the Neurogenic Bowel Dysfunction Scale | Baseline (Week 0), Week 4, and Week 12
  Neurogenic bowel dysfunction will be assessed using the Neurogenic Bowel Dysfunction (NBD) Scale, a validated questionnaire for individuals with spinal cord injury.
  The scale ranges from 0 to 47 points, with higher scores indicating more severe bowel dysfunction.
  The outcome measure is the change in total NBD score from baseline (Week 0) to Week 12.
Change in Bowel Care Time Measured in Minutes | Baseline (Week 0), Week 4, and Week 12
  Bowel care time will be measured as the average time (in minutes) required to complete bowel care management.
  Time will be self-reported by participants. The outcome measure is the change in bowel care time from baseline (Week 0) to Week 12.

SECONDARY OUTCOMES:
Change in Fecal Incontinence Rate | Baseline (Week 0), Week 4, and Week 12
  Fecal incontinence will be assessed based on self-reported occurrence of fecal incontinence episodes.
  The outcome will be expressed as the percentage of participants experiencing fecal incontinence at baseline (Week 0), Week 4, and Week 12.

IPD SHARING:
Plan to Share IPD: No
As the process cannot be anticipated, no plan has been established.